CLINICAL TRIAL: NCT02549053
Title: Prevalence of Human Papillomavirus in Barrett Esophagus Compared With Controls
Acronym: Barrett
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CP 2011-10
Record Dates: First submitted 2015-07-30; First posted 2015-09-14 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Barrett esophagus patients (Experimental): esophagus biopsies (pathologic and healthy zones)
  Interventions: Procedure: esophagus biopsies (pathologic and healthy zones)
- control patients (Sham Comparator): esophagus biopsies (healthy zones)
  Interventions: Procedure: esophagus biopsies (healthy zones)

INTERVENTIONS:
Procedure: esophagus biopsies (pathologic and healthy zones) — Biopsies were realised in the distal third of esophagus : 4 for Barrett esophagus patients (2 in healthy zone, 2 in pathological zone).
  Arms: Barrett esophagus patients
Procedure: esophagus biopsies (healthy zones) — Biopsies were realised in the distal third of esophagus :2 for control patients in healthy zone
  Arms: control patients

SUMMARY:
The aim of this study was to determine whether the prevalence of Human PapillomaVirus (HPV) was increased in patients with Barrett esophagus compared with controls in a prospective study. Secondary objective was to identify, if present, the type of Human PapillomaVirus (HPV) associated in Barrett esophagus.

DETAILED DESCRIPTION:
Barrett's esophagus (BE) is defined by the replacement of normal stratified squamous epithelium in the distal third of esophagus by specialized intestinal metaplasia. It is related to gastro-esophageal reflux disease. Diagnosis is suspected during endoscopy and confirmed on biopsy. The classification of CM from Prague is validated to describe BE during endoscopy. The main complication of the BE is adenocarcinoma, according to metaplasia-dysplasia-cancer sequence. The incidence of esophageal adenocarcinoma is variable, ranging from 0.4 to 3 %. BE is found in 100% esophageal adenocarcinoma and in 42% junction adenocarcinoma. Among the unknown risk factors involved in the onset of dysplasia, viruses can't be excluded.

It is well established that Human Papillomavirus (HPV) is strongly associated with squamous cell dysplasia of female uterine cervix and its progression to cervical carcinoma. HPV is also implicated in others invasive carcinomas including uterine cervix, vulvar, vaginal, anal, penile, head and neck squamous cell carcinoma. Several studies showed that HPV could be associated in head and neck cancers and that tumor HPV status in patients with oropharyngeal squamous cell carcinomas was an independent prognostic factor for survival. The association between HPV and esophageal squamous cell carcinomas is still controversed with epidemiological studies reporting prevalence of mucosal HPV DNA ranging from 0 to 70%. Studies that have investigated HPV and adenocarcinoma of esophagus or Barrett's esophagus (BE) are scarce and data are not clear. A recent prospective study showed that HPV was strongly associated with Barrett'dysplasia and esophageal adenocarcinoma.

The aim of this study was to determine whether the prevalence of HPV was increased in patients with BE compared with controls in a prospective study. Secondary objective was to identify, if present, the type of HPV associated in BE.

ELIGIBILITY:
Inclusion Criteria:

* written consent obtained before gastroscopy,
* patients aged more than 18 years,
* normal coagulation parameters Inclusion criteria for group A "control" and B "BE" were as follows, respectively: patients undergoing gastroscopy for non esophageal reason and presented no clinical, endoscopic or histopathological evidence of GERD or complication and patients undergoing gastroscopy for BE surveillance or suspected BE during gastroscopy.

Exclusion Criteria:

* written consent not obtained before gastroscopy,
* inability to give informed consent,
* pregnant or nursing women,
* major person protected by french law,
* person who is not affiliated to a social security regime,
* patient who is in a exclusion period for another clinical study,
* curative anticoagulation treatment,
* hemostatic disturbances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2012-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Research of HPV DNA in esophagus biopsies using real time polymerase chain reaction (PCR) | up to 14 months, time to develop analysis technique at the virology lab, then to collect enough biopsies to start analysis phase
  Research of HPV DNA using real time polymerase chain reaction (PCR)

CONTACTS AND LOCATIONS:
Overall Officials: François-Xavier Caroli-Bosc, PhD, Principal Investigator — UH Angers
Locations (2):
- France (2):
  - UH Angers, Angers
  - UH Nantes, Nantes

REFERENCES:
- [Derived] Brochard C, Ducancelle A, Pivert A, Bodin M, Ricard A, Coron E, Couffon C, Dib N, Luet D, Musquer N, Rhun ML, Bertrais S, Michalak S, Lunel-Fabiani F, Cesbron-Metivier E, Caroli-Bosc FX. Human papillomavirus does not play a role in the Barrett esophagus: a French cohort. Dis Esophagus. 2017 Nov 1;30(11):1-7. doi: 10.1093/dote/dox088. PMID 28881904